CLINICAL TRIAL: NCT04642430
Title: COmparison of Bleeding Risk Between Rivaroxaban and Apixaban in Patients With Atrial Fibrillation
Acronym: COBRRA-AF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Venous Thromboembolism Clinical Trials and Outcomes Research (CanVECTOR) Network (Network); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COBRRA-AF
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation
Keywords: Stroke Prevention; Bleed
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage | interventions — apixaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: A pragmatic prospective randomized open blinded endpoint (PROBE) trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban group (Active Comparator): 5 mg PO, twice daily for 12 months of treatment. A dose reduction* to 2.5 mg twice daily will apply if patients meet 2 of 3 following criteria: age > 80 years; weight < 60 kg; creatinine >133 micromol/L.
  *Patients with AF who are receiving DOAC should have their renal function assessed at baseline and at least annually
  Interventions: Drug: Apixaban
- Rivaroxaban Group (Active Comparator): 20 mg PO, once daily for 12 months of treatment. A dose reduction* to 15 mg daily will apply to patients with creatinine clearance <50 ml/min.
  *Patients with AF who are receiving DOAC should have their renal function assessed at baseline and at least annually
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Apixaban — Refer to Apixaban group
  Other Names: Eliquis
  Arms: Apixaban group
Drug: Rivaroxaban — Refer to Rivaroxaban group
  Other Names: Xarelto
  Arms: Rivaroxaban Group

SUMMARY:
Atrial Fibrillation (AF) affects 200,000 Canadians and increases risk of stroke, morbidity and mortality. Having a stroke can affect a patient's ability to speak, eat, walk, work, care for themselves, and interact with others. Not only can it ruin one's life, but it can also be fatal. A stroke occurs when blood flow to the brain is blocked by a clot, depriving brain cells of oxygen. In people with atrial fibrillation, blood flow is sluggish in the top chambers of the heart, and blood clots can form there. When a piece of a clot breaks off, it can travel to the brain and cause a stroke. That's where blood thinners come in. Blood thinners, or anticoagulants, decrease the chances of blood clots forming in the heart, reducing the risk of stroke. Studies show that blood thinners are highly effective at reducing the risk of stroke by up to 95%.

The conventional blood thinner is warfarin, taken by mouth. Warfarin requires regular blood tests to make sure a patient getting the correct dose. The patient also may have to avoid certain foods since the medication can interact with them. Newer blood thinners, known as direct-oral anticoagulants (DOACs) are available, which do not require regular blood tests and do not interact with foods. Two of the new blood thinners are called rivaroxaban and apixaban. Like warfarin, they can be taken by mouth, and studies have shown them to be as effective as warfarin.

Both rivaroxaban and apixaban have been approved for stroke prevention in AF by Health Canada. However, there have been no direct head-to-head comparisons of these two anticoagulants, meaning comparative safety data is not available. Increasing use of DOACs for stroke prevention in AF and patient values around bleeding highlight the need for a comparison trial to ensure patients receive the anticoagulant with the greatest balance of benefit to potential harm.

The trial is to assess bleeding rates and superiority of using apixaban versus rivaroxaban in patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) affects 200,000 Canadians and increases risk of stroke, morbidity and mortality. Oral anticoagulants such as Vitamin K antagonists (VKAs) and direct oral anticoagulants (DOACs) are highly effective at reducing the risk of stroke by up to 95%. Randomized controlled trials (RCTs) have compared apixaban and rivaroxaban (both DOACs) to VKAs for stroke prevention in AF, and are approved for this use by Health Canada. However, there have been no direct head-to-head comparisons of these two anticoagulants, meaning comparative safety data is not available. Increasing use of DOACs for stroke prevention in AF, patient values around bleeding, and litigation highlight the need for a comparison trial to ensure patients receive the anticoagulant with the greatest balance of benefit to potential harm.

The objective of this RCT is to compare the safety of the first 12 months of apixaban twice daily to rivaroxaban once daily in patients with non-valvular AF (NVAF). Patients will be monitored for the primary outcome of clinically relevant bleeding (CRB; a composite of major bleeding (MB) and clinically relevant non-major bleeding (CRNMB) events during follow-up. This trial will directly inform clinical practice and the choice of first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Confirmed new diagnosis of AF on ECG with an indication to start anticoagulation according to Canadian Cardiovascular Society guidelines

Exclusion Criteria:

* Creatinine clearance =<15 ml/min calculated using the Cockcroft-Gault formula
* Any contraindication for anticoagulation with apixaban or rivaroxaban as determined by the treating physician such as, but not limited to:

  * active bleeding
  * history of mechanical valve
  * other indication for anticoagulation (e.g. mechanical valves, venous thrombosis)
  * dual antiplatelet agent use
  * known liver disease with coagulopathy
  * use of contraindicated medications (strong inducers/inhibitors of CYP 3A4/5, P-glycoprotein)
  * pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3018 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of adjudicated clinically relevant bleeding (CRB) events | For the duration of the study: 12 months
  CRB events are defined as the composite of major bleeding (MB) events and clinically relevant non-major bleeding (CRNMB) events

SECONDARY OUTCOMES:
Adjudicated Major Bleeding events | For the duration of the study: 12 months
  Major Bleeding includes clinically overt bleeding and is associated with:
  * Fatal bleeding, and/or
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
  * A fall in hemoglobin of ≥20 g/L, or
  * Leading to transfusion of ≥2 units of whole blood or red cells.
Adjudicated Clinically Relevant Non-Major Bleeding events | For the duration of the study: 12 months
  Clinically relevant non-major bleeding will be defined as:
  • Any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  * Requiring medical intervention by a healthcare professional
  * Leading to hospitalization or increased level of care
  * Prompting a face to face (i.e., not just a telephone or electronic communication) evaluation
Adjudicated stroke/TIA events | For the duration of the study: 12 months
  Stroke is defined as non-traumatic focal neurologic deficit lasting ≥ 24 hours and confirmed on cerebral imaging (computed tomography or magnetic resonance imaging).
  Transient ischemic attack (TIA) is defined as a temporary loss of blood flow to a part of the brain with focal neurologic deficit lasting < 24 hours without imaging evidence of acute infarction.
  Strokes are to be classified as ischemic, hemorrhagic stroke, or uncertain. Hemorrhagic strokes are considered and will be reported as both bleeding events as well as stroke endpoints. The location of the bleeding can be determined from the diagnostic imaging reports.
All-cause mortality | For the duration of the study: 12 months
  Using a binary outcome of an event or no event (Individual rates of death, all causes).
Medication adherence | For the duration of the study: 12 months
  Reported as the number of patients self-reporting "all assigned medications were taken" "missing at least one dose of study medication", or "not able to take all of the study medications" out of the total number of medication compliance assessments done respectively
Incremental cost-effectiveness ratio | For the duration of the study: 12 months
  We will model the prognosis of a cohort of patients receiving rivaroxaban versus apixaban. The results will be presented as incremental cost per QALY gained, incremental costs per one clinically relevant bleeding cases prevented, and incremental cost per one life year saved.

CONTACTS AND LOCATIONS:
Overall Officials: Lana Castellucci, MD, FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (8):
- Canada (8):
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - University Ottawa Heart Institute, Ottawa, Ontario
  - CISSS de l'Outaouais, Gatineau, Quebec
  - CHU de Quebec - Université Laval, Laval, Quebec
  - Ciusss Nim, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No